CLINICAL TRIAL: NCT01309841
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of NKTR-118 in Patients With Non-Cancer-Related Pain and Opioid-Induced Constipation (OIC)
Brief Title: Assessment of Efficacy and Safety in Patients With Non-cancer-related Pain and Opioid-induced Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3820C00004; 2011-001987-24 (EudraCT Number)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Induced Constipation (OIC)
Keywords: Non-Cancer-Related Pain, Opioid-Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Oral treatment
  Interventions: Drug: NKTR-118
- 2 (Experimental): Oral treatment
  Interventions: Drug: NKTR-118
- 3 (Placebo Comparator): Oral treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NKTR-118 — 12.5 mg oral tablet once daily
  Arms: 1
Drug: NKTR-118 — 25 mg oral tablet once daily
  Arms: 2
Drug: Placebo — Oral tablet once daily
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the effect and safety of NKTR-118 treatment of opioid-induced constipation in patients with non-cancer-related pain, including those patients that have inadequate response to laxative therapy (LIR).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study-specific procedures.
* Men and women who are between the ages of ≥18 and <85 years.
* Self-reported active symptoms of OIC at screening (<3 SBMs/week and experiencing ≥1 reported symptom of hard/lumpy stools, straining, or sensation of incomplete evacuation/anorectal obstruction in at least 25% of BMs over the previous 4 weeks); and Documented confirmed OIC (<3 SBMs/week on average over the 2-week OIC confirmation period.
* Receiving a stable maintenance opioid regimen consisting of a total daily dose of 30 mg to 1000 mg of oral morphine, or equianalgesic amount(s) of 1 or more other opioid therapies for a minimum of 4 weeks prior to screening for non-cancer-related pain with no anticipated change in opioid dose requirement over the proposed study period as a result of disease progression.
* Willingness to stop all laxatives and other bowel regimens including prune juice and herbal products throughout the 2-week OIC confirmation period and the 12-week treatment period, and to use only bisacodyl as rescue medication if a BM has not occurred within at least 72 hours of the last recorded BM.

Exclusion Criteria:

* Patients receiving Opioid regimen for treatment of pain related to cancer.
* History of cancer within 5 years from first study visit with the exception of basal cell cancer and squamous cell skin cancer.
* Medical conditions and treatments associated with diarrhea, intermittent loose stools, or constipation.
* Other issues to the gastrointestinal tract that could impose a risk to the patient.
* Pregnancy or lactation.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, Study Director — AstraZeneca Pharmaceuticals, Wilm DE
Locations (117):
- United States (91):
  - Research Site, Birmingham, Alabama
  - Research Site, Calera, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Malvern, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site, Garden Grove, California
  - Research Site, Laguana Hills, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, Los Gatos, California
  - Research Site, Montebello, California
  - Research Site, National City, California
  - Research Site, Norwalk, California
  - Research Site, Paramount, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Denver, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, Brooksville, Florida
  - Research Site, DeLand, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jackson, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Plantation, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Venice, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Bloomington, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Greenfield, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Pikesville, Maryland
  - Research Site, Brockton, Massachusetts
  - Research Site, Kalamazoo, Michigan
  - Research Site, Biloxi, Mississippi
  - Research Site, Saint Joseph, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Trenton, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Morrisville, North Carolina
  - Research Site, Beavercreek, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Medord, Oregon
  - Research Site, Feasterville, Pennsylvania
  - Research Site, Huntingdon Valley, Pennsylvania
  - Research Site, Levittown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Yardley, Pennsylvania
  - Research Site, Cumberland, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Clarksville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Doral, Texas
  - Research Site, Houston, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Spokane, Washington
- Australia (8):
  - Research Site, Broadmeadow, New South Wales
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Port Kembla, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Greenslopes, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Fremantle, Western Australia
  - Research Site, Nedlands, Western Australia
- Germany (14):
  - Research Site, Potsdam, BR
  - Research Site, Hamburg, Hamburg
  - Research Site, Dietzenbach, Hesse
  - Research Site, Hüttenberg, Hesse
  - Research Site, Wetzlar, Hesse
  - Research Site, Celle, Lower Saxony
  - Research Site, Hanover, Lower Saxony
  - Research Site, Schwerin, Mecklenburg-Vorpommern
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Mainz, Rhineland-Palatinate
  - Research Site, Dresden, Saxony
  - Research Site, Leipzig, Saxony
  - Research Site, Kiel, Schleswig-Holstein
  - Research Site, Berlin, State of Berlin
- Slovakia (4):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Prešov

REFERENCES:
- [Derived] Webster L, Tummala R, Diva U, Lappalainen J. A 12-week extension study to assess the safety and tolerability of naloxegol in patients with noncancer pain and opioid-induced constipation. J Opioid Manag. 2016 Nov/Dec;12(6):405-419. doi: 10.5055/jom.2016.0360. PMID 28059433
- [Derived] Lawson R, King F, Marsh K, Altincatal A, Cimen A. Impact of Treatment with Naloxegol for Opioid-Induced Constipation on Patients' Health State Utility. Adv Ther. 2016 Aug;33(8):1331-46. doi: 10.1007/s12325-016-0365-y. Epub 2016 Jun 24. PMID 27342744
- [Derived] Tack J, Lappalainen J, Diva U, Tummala R, Sostek M. Efficacy and safety of naloxegol in patients with opioid-induced constipation and laxative-inadequate response. United European Gastroenterol J. 2015 Oct;3(5):471-80. doi: 10.1177/2050640615604543. PMID 26535126
- [Derived] Chey WD, Webster L, Sostek M, Lappalainen J, Barker PN, Tack J. Naloxegol for opioid-induced constipation in patients with noncancer pain. N Engl J Med. 2014 Jun 19;370(25):2387-96. doi: 10.1056/NEJMoa1310246. Epub 2014 Jun 4. PMID 24896818
- See also: Clinical_Study_Report_Synopsis_D3820C00004 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1853&filename=Clinical_Study_Report_Synopsis_D3820C00004.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in Australia, Germany, Slovakia, and the United States between 14 March 2011 and 16 August 2012.
Pre-assignment Details: The study duration was up to 18 weeks, consisting of an initial screening period lasting up to 2 weeks, a 2-week OIC confirmation period, during which the diagnosis of OIC and stability of the opioid regimen were confirmed, a 12-week treatment period, and a follow-up visit 2 weeks after the last dose of study drug.
Groups:
- NKTR-118 12.5 mg: NKTR-118 12.5 QD, oral treatment
- NKTR-118 25 mg: NKTR-118 25 mg QD, oral treatment
- Placebo: Placebo QD, oral treatment
Period: Overall Study
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Started | 217 | 218 | 217
Completed | 178 | 177 | 180
Not Completed | 39 | 41 | 37
Not completed — Other | 0 | 1 | 1
Not completed — Lost to Follow-up | 7 | 6 | 4
Not completed — Study-Specific Withdrawal Criteria | 3 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Adverse Event | 9 | 22 | 11
Not completed — Death | 1 | 0 | 0
Not completed — Eligibility Criteria Not Fulfilled | 0 | 0 | 1
Not completed — Withdrawal by Subject | 17 | 6 | 13
Not completed — Did Not Receive Treatment | 2 | 0 | 1
Not completed — Severe non-compliance with protocol | 0 | 5 | 2

BASELINE CHARACTERISTICS:
Population: A total of 11 patients (4 patients each in the NKTR-118 25 mg and 12.5 mg groups and 3 patients in the placebo group) had been previously randomized within the NKTR-118 program at a different study center. These patients were excluded from the ITT and Safety analysis sets. Baseline characteristics are summarized based on the ITT analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo | Total
Number analyzed (Participants) | 213 | 214 | 214 | 641
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (10.43) | 52.2 (10.29) | 52.9 (9.99) | 52.3 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 118 | 140 | 393
  Male | 78 | 96 | 74 | 248
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 5 | 1 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 42 | 38 | 44 | 124
  White | 164 | 173 | 160 | 497
  Other | 1 | 2 | 4 | 7
Baseline laxative response status [Number; unit: Participants] — Laxative response status was determined at the screening visit (Visit 1) based on the Baseline Laxative Response Status Questionnaire. Patients were classified as: Laxative Inadequate Responder (LIR: patients who reported moderate, severe, or very severe symptoms in at least 1 of the 4 stool symptom domains); Laxative Adequate Responder (LAR: patients who reported no symptoms or only mild symptoms); and Laxative Unknown Responder (LUR: patients who had not taken laxatives over the previous 2 weeks or who had taken 1 or more laxative classes on <4 days over the previous 2 weeks).
  Participants
    Laxative Inadequate Response (LIR) | 115 | 117 | 118 | 350
    Laxative Adequate Response (LAR) | 3 | 2 | 2 | 7
    Laxative Unknown Response (LUR) | 95 | 95 | 94 | 284

OUTCOME MEASURES:

1. Primary Outcome: Response (Responder/Non-responder) to Study Drug During Weeks 1 to 12
Description: Responder was defined as having at least 3 spontaneous bowel movements (SBMs)/week with at least 1 SBM/week increase over baseline for at least 9 out of the 12 treatment weeks and 3 out of the last 4 treatment weeks during the double-blind treatment period. An SBM is a bowel movement occurring 24 hours or more since the last use of rescue medication.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: The ITT analysis set included all randomized patients, with the exception of patients who were found to have randomized multiple times within the program at different centers.
Measure: Number; unit: Number of patients
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 213 | 214 | 214
Number of patients | 87 | 95 | 63
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; Analysis via Cochran Mantel-Haenszel test stratified by response to laxatives at baseline (LIR, LAR, LUR); Test type: Superiority or Other; p = 0.015, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.380, 95% CI 2-sided [1.062 to 1.795]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; Analysis via Cochran Mantel-Haenszel test stratified by response to laxatives at baseline (LIR, LAR, LUR); Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.509, 95% CI 2-sided [1.168 to 1.949]

2. Secondary Outcome: Response (Responder/Non-responder) to Study Drug in the LIR Subgroup During Weeks 1 to 12
Description: Responder is defined as having at least 3 SBMs/week, with at least 1 SBM/week increase over baseline for at least 9 out of 12 weeks and at least 3 out of the last 4 weeks.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: The ITT analysis set included all randomized patients, with the exception of patients who were found to have randomized multiple times within the program at different centers. The LIR subgroup used 1 or more laxative classes for at least 4 days in the 2 weeks prior to entry and reported moderate to very severe symptoms.
Measure: Number; unit: Number of patients
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 115 | 117 | 118
Number of patients | 49 | 57 | 34
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; Test type: Superiority or Other; p = 0.028, Cochran-Mantel-Haenszel — Response rate over Weeks 1 to 12 in the LIR subgroup is a key secondary endpoint included in the multiple testing procedure; Risk Ratio (RR) = 1.479, 95% CI 2-sided [1.038 to 2.107]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.691, 95% CI 2-sided [1.205 to 2.373]

3. Secondary Outcome: Time (in Hours) to First Post-dose Laxation Without the Use of Rescue Laxatives Within the Previous 24 Hours
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 213 | 214 | 214
Hours | 20.4 [11.5 to 22.7] | 5.9 [4.8 to 11.5] | 35.8 [27.0 to 48.1]

4. Secondary Outcome: Change From Baseline in Mean Number of Days Per Week With at Least 1 SBM During Weeks 1 to 12
Time Frame: 12 weeks
Population: The ITT analysis set included all randomized patients who had evaluable data at baseline and post-baseline, with the exception of patients who were found to have randomized multiple times within the program at different centers.
Measure: Least Squares Mean (Standard Error); unit: Number of Days
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 211 | 212 | 211
Number of Days | 2.21 (0.13) | 2.48 (0.13) | 1.66 (0.13)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; Analysis via Mixed Model Repeated Measures (MMRM) with fixed effects for baseline, baseline laxative response, treatment and treatment time interaction. Study pooled center is included as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 0.55, 95% CI 2-sided [0.24 to 0.86]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; Analysis via MMRM with fixed effects for baseline, baseline laxative response, treatment and treatment time interaction. Study pooled center is included as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Ls mean difference = 0.82, 95% CI 2-sided [0.51 to 1.13]

5. Secondary Outcome: Change From Baseline in Degree of Straining
Description: A single-item straining question was asked via the eDiary: "How much did you strain during your bowel movement?" Patients responded on a 5 point Likert scale: 1=Not at all; 2=A little bit; 3=A moderate amount; 4=A great deal; 5=An extreme amount. A negative change from baseline indicates improvement.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 211 | 212 | 211
units on a scale | -0.64 (0.05) | -0.73 (0.05) | -0.54 (0.05)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; Analysis via MMRM with fixed effects for baseline, baseline laxative response (LIR, non-LIR), treatment and treatment time interaction. Study pooled center is included as a random effect; Test type: Superiority or Other; p = 0.176, Mixed Models Analysis; LS mean difference = -0.09, 95% CI 2-sided [-0.23 to 0.04]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; LS mean difference = -0.18, 95% CI 2-sided [-0.32 to -0.05]

6. Secondary Outcome: Change From Baseline in Stool Consistency (Bristol Stool Scale)
Description: Patients rated stool consistency through completion of the BSS after each BM. The 7 stool types are: 1. Separate hard lumps, like nuts (hard to pass); 2. Sausage-shaped, but lumpy; 3. Like sausage, but with cracks on its surface; 4. Like a sausage or snake, smooth and soft; 5. Soft blobs with clear cut edges (passed easily); 6. Fluffy pieces with ragged edges, a mushy stool; 7. Watery, no solid pieces. A positive change from baseline indicates improvement.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 211 | 212 | 211
units on a scale | 0.53 (0.07) | 0.66 (0.07) | 0.47 (0.07)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.564, Mixed Models Analysis; LS mean difference = 0.05, 95% CI 2-sided [-0.12 to 0.23]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.042, Mixed Models Analysis; LS mean difference = 0.18, 95% CI 2-sided [0.01 to 0.36]

7. Secondary Outcome: Change From Baseline in Percent Numbers of Days With a CSBM (Complete Spontaneous Bowel Movement)
Description: A single-item question on the completeness of evacuation, developed and validated through 1:1 interviews with OIC patients, was asked via the eDiary: "Did you feel like your bowels were completely empty after the bowel movement?" Patients provided a yes or a no response. A positive change from baseline indicates improvement.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent days/week
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 211 | 212 | 211
Percent days/week | 22.31 (1.73) | 27.04 (1.75) | 18.45 (1.72)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.094, Mixed Models Analysis; LS mean difference = 3.87, 95% CI 2-sided [-0.66 to 8.39]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 8.59, 95% CI 2-sided [4.04 to 13.14]

8. Secondary Outcome: Change From Baseline in Mean Spontaneous Bowel Movements/Week
Description: The number of spontaneous bowel movements/week was determined from the patient's eDiary.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Number of SBMs/week
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 211 | 212 | 211
Number of SBMs/week | 2.56 (0.18) | 3.02 (0.18) | 2.02 (0.18)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis; LS mean difference = 0.54, 95% CI 2-sided [0.12 to 0.96]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 0.99, 95% CI 2-sided [0.57 to 1.41]

9. Secondary Outcome: Time (in Hours) to First Post-dose Laxation Without the Use of Rescue Laxatives Within the Previous 24 Hours in the Laxative Inadequate Response (LIR) Subgroup
Description: Time to first post-dose laxation without the use of rescue laxatives within the last 24 hours was calculated in hours as: Date/Time of first post-dose laxation without rescue - First dose date/time.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 115 | 117 | 118
hours | 20.6 [8.1 to 23.5] | 5.4 [3.9 to 10.7] | 43.4 [25.2 to 48.2]

10. Secondary Outcome: Change From Baseline in Patient Assessment of Constipation Symptoms Questionnaire (PAC-SYM)
Description: The PAC-SYM questionnaire is a 12-item questionnaire that evaluates the severity of symptoms of constipation in 3 domains (stool, rectal, and abdominal symptoms) on a 5-point Likert scale ranging from 0 (absent) to 4 (very severe) in the 2 weeks (14 days) prior to assessment. Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items (ie, symptoms). The range of the domain or total score is 0 (response is 'absent' for each item) to 4 (response is 'very severe' for each item). A negative change from baseline indicates improvement.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: The ITT analysis set included all randomized patients who had evaluable data at baseline and post-baseline, with the exception of patients who randomized multiple times at different centers. MMRM analysis includes all patients with baseline and at least 1 post-baseline assessment, while the Ns at Week 12 reflect patients providing data at Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 171 | 158 | 173
units on a scale
  Total score | -0.76 (0.05) | -0.81 (0.05) | -0.69 (0.05)
  Abdominal symptoms subscore | -0.61 (0.06) | -0.65 (0.06) | -0.63 (0.06)
  Rectal symptoms subscore | -0.66 (0.05) | -0.73 (0.05) | -0.53 (0.05)
  Stool symptoms subscore | -0.96 (0.07) | -1.00 (0.07) | -0.84 (0.07)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.273, Mixed Models Analysis — Analysis for change in PAC-SYM total score from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.08, 95% CI 2-sided [-0.21 to 0.06]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.089, Mixed Models Analysis — Analysis for change in PAC-SYM total score from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.12, 95% CI 2-sided [-0.26 to 0.02]
Statistical Analysis 3: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.849, Mixed Models Analysis — Analysis for change in PAC-SYM abdominal symptoms subscore from baseline (Week 1) to end of treatment (Week 12); Slope = 0.02, 95% CI 2-sided [-0.14 to 0.17]
Statistical Analysis 4: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.749, Mixed Models Analysis — Analysis for change in PAC-SYM abdominal symptoms subscore from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.03, 95% CI 2-sided [-0.18 to 0.13]
Statistical Analysis 5: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.062, Mixed Models Analysis — Analysis for change in PAC-SYM rectal symptoms subscore from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.13, 95% CI 2-sided [-0.26 to 0.01]
Statistical Analysis 6: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — Analysis for change in PAC-SYM rectal symptoms subscore from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.21, 95% CI 2-sided [-0.35 to -0.07]
Statistical Analysis 7: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.202, Mixed Models Analysis — Analysis for change in PAC-SYM stool symptoms subscore from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.11, 95% CI 2-sided [-0.29 to 0.06]
Statistical Analysis 8: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.072, Mixed Models Analysis — Analysis for change in PAC-SYM stool symptoms subscore from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.16, 95% CI 2-sided [-0.34 to 0.01]

11. Secondary Outcome: Change From Baseline in Patient Assessment of Constipation Quality of Life (PAC-QOL) Satisfaction Domain
Description: The PAC-QOL scale is a 28-item self-report instrument designed to evaluate the burden of constipation on patients' everyday functioning and well-being in the 2 weeks (14 days) prior to assessment. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). The instrument can be used to generate an overall score, but is also reported to assess 4 specific constipation-related domains including: 1) Worries and concerns (11 items), 2) Physical discomfort (4 items), 3) Psychosocial discomfort (8 items), and 4) Satisfaction (5 items). Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items. The range of the domain or total score is 0 (response is 'not at all' for each item) to 4 (response is 'extremely' for each item). A negative change from baseline indicates improvement.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 172 | 159 | 174
units on a scale | -0.91 (0.09) | -1.06 (0.09) | -0.89 (0.09)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; Analysis via MMRM with fixed effects for baseline, baseline laxative response, treatment and treatment time interaction. Due to convergence issues, study pooled center is also included as a fixed, rather than random effect; Test type: Superiority or Other; p = 0.831, Mixed Models Analysis; LS mean difference = -0.02, 95% CI 2-sided [-0.25 to 0.20]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.141, Mixed Models Analysis; LS mean difference = -0.18, 95% CI 2-sided [-0.41 to 0.06]

ADVERSE EVENTS:
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 11/211 | 7/214 | 11/213
Other Adverse Events (participants affected / at risk) | 57/211 | 85/214 | 53/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 12.5 mg (N=211) | NKTR-118 25 mg (N=214) | Placebo (N=213)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
SIGMOIDITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 2 (2) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CARDIAC VALVE REPLACEMENT COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
TENDON INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RENAL CANCER STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BASILAR MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 12.5 mg (N=211) | NKTR-118 25 mg (N=214) | Placebo (N=213)
ABDOMINAL PAIN (Gastrointestinal disorders) | 19 (21) | 26 (28) | 7 (8)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (3) | 11 (13) | 4 (5)
DIARRHOEA (Gastrointestinal disorders) | 7 (8) | 19 (20) | 9 (9)
FLATULENCE (Gastrointestinal disorders) | 8 (8) | 12 (12) | 5 (5)
NAUSEA (Gastrointestinal disorders) | 16 (19) | 16 (19) | 10 (10)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 7 (7) | 5 (5) | 4 (4)
VOMITING (Gastrointestinal disorders) | 4 (4) | 7 (12) | 7 (7)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (6) | 8 (8) | 7 (7)
URINARY TRACT INFECTION (Infections and infestations) | 5 (6) | 0 (0) | 6 (6)
FALL (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 6 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8) | 5 (5)
DIZZINESS (Nervous system disorders) | 3 (4) | 0 (0) | 5 (5)
HEADACHE (Nervous system disorders) | 5 (5) | 8 (8) | 4 (4)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days